CLINICAL TRIAL: NCT05291663
Title: Retrospective Study of Effect of Accelerated Radiation Therapy , Six Fractions Per Week , for Squamous Cell Carcinoma of Head and Neck.
Brief Title: Effect of Accelerated RTH in Squamous Cell Carcinoma in Head and Neck
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zienab Kamel Mahmoud, Doctor, Assiut University
Other Study IDs: RTH in head & neck tumors
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the efficacy of the accelerated radiotherapy in squamous cell carcinoma of head and neck

DETAILED DESCRIPTION:
* HNSCC is the sixth most common cancer worldwide, with 890.000 new cases and 450.000 deaths in 2018.
* The incidence of HNSCC continues to rise and is anticipated to increase by 30% (that is, 1.08 million new cases annually) by 2030.
* Squamous cell carcinoma constitutes 90% of all head and neck cancers and it predominates in males.
* Risk factors such as cigarette consumption and alcohol consumption, are well established.
* Treatment decisions are guided by clinic-pathologic factors such as age and stage.
* Treatment of the majority of patients with HNSCC requires multimodality approaches.
* Radiotherapy or surgery alone can be considered as the standard treatment modality for patients having early head and neck squamous cell carcinoma.
* When conventionally fractionated radiotherapy is used, long-term tumor control can be achieved in less than 30% of patients with advanced head and neck carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients of (18 up to 75 years of age)
* Performance status of 0-2 according to ECOG scale.
* Patients with no prior chemotherapy, radiotherapy or surgery except for biopsy.

Exclusion Criteria:

* Patients with previous irradiation to head and neck.
* Pregnant or lactating women.
* Patients with impaired heart or lung diseases.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: -Patients of (18 up to 75 years of age)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Determine progression-free survival rate | Baseline
  Determine the toxicity and loco-regional control by using accelerated RTH in squamous cell carcinoma in head and neck

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa El-sayed Abd Elwanis, Study Director — Assiut University

REFERENCES:
- [Result] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Result] Windon MJ, D'Souza G, Rettig EM, Westra WH, van Zante A, Wang SJ, Ryan WR, Mydlarz WK, Ha PK, Miles BA, Koch W, Gourin C, Eisele DW, Fakhry C. Increasing prevalence of human papillomavirus-positive oropharyngeal cancers among older adults. Cancer. 2018 Jul 15;124(14):2993-2999. doi: 10.1002/cncr.31385. Epub 2018 Apr 30. PMID 29710393
- [Result] Blot WJ, McLaughlin JK, Winn DM, Austin DF, Greenberg RS, Preston-Martin S, Bernstein L, Schoenberg JB, Stemhagen A, Fraumeni JF Jr. Smoking and drinking in relation to oral and pharyngeal cancer. Cancer Res. 1988 Jun 1;48(11):3282-7. PMID 3365707
- [Result] Johnson DE, Burtness B, Leemans CR, Lui VWY, Bauman JE, Grandis JR. Head and neck squamous cell carcinoma. Nat Rev Dis Primers. 2020 Nov 26;6(1):92. doi: 10.1038/s41572-020-00224-3. PMID 33243986